CLINICAL TRIAL: NCT05397964
Title: Retrospective Evaluation of the Results of Direct Pulp Capping Treatment
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Funda Ozturk Bozkurt, Assosciate Professor, Istanbul Medipol University Hospital
Other Study IDs: 362
Record Dates: First submitted 2022-05-11; First posted 2022-05-31 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Pulp Exposure, Dental
Keywords: direct pulp capping,; calcium hydroxide liner
MeSH Terms: conditions — Dental Pulp Exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Radiopaque Calcium Hydroxide Composition — Treatment of exposed pulp tissue with radiopaque calcium hydroxide composition as a direct pulp capping material

SUMMARY:
The aim of this retrospective study is to evaluate the vitality of teeth that had been treated with calcium hydroxide in direct pulp capping cases.

DETAILED DESCRIPTION:
During restorative procedures, pulp tissue may be exposed while caries is removed from deep dentin tissue. There are some defense mechanisms to protect against bacterial invasion, but the best barrier is provided by living pulp tissue. During the life of a tooth, living pulp tissue is responsible for the formation of secondary dentin, peritubular dentin, and repair dentin in response to biological or pathological stimuli. Direct pulp capping means closing the exposed pulp tissue with the aim of healing. Calcium hydroxide, a biocompatible material, has been used for many years in pulp capping, with its ability to reduce bacterial infection and promote dentinopulpal remineralization. However, the results regarding the long-term clinical success of direct pulp capping with calcium hydroxide are conflicting. After the calcium hydroxide application, the restoration should be done with a filling material that can prevent the bacteria transfer between the restoration and the tooth tissue in the long term. The success of the restoration has a significant impact on the healing and treatment outcome. The aim of this study is to evaluate the clinical success of 217 direct capping treatments and restorations ,which were routinely applied to 190 patients in our clinic between 2011 and 2020.

Individuals who were invited to the control session and approved to participate in the research with their signatures, to evaluate the result of direct capping treatment, will be examined by:

* Visual examination: Related teeth and soft tissue will be examined.
* Palpation: The apex of the related tooth will be palpated intra and extra orally.
* Percussion: Percussion will be performed on the related tooth horizontally and vertically with a handpiece.
* Cold test: Ethyl chloride (Chloraethyl, IGS AEROSOLS GMBH, Baden, Germany) cold spray is applied to a small cotton pellet to the symmetrical tooth, which is thought to be alive, for control purposes, and then to the cervical 1/3 of the relevant tooth for 2-3 seconds.Sensitivity will be asked. A sensitive tooth will be considered to have responded positively to the cold test. In the absence of sensitivity, the tooth will be considered to have given a negative response.
* Electric pulp test: For control purposes, first the symmetrical tooth, which is thought to be alive, and then the related tooth will be tested with the Digitest Pulp Vitality Tester (Parkell, INC., New York, USA). Before the test, the teeth will be isolated from saliva with a cotton pad and toothpaste will be used as a conductive. During the application, the patient will be asked whether she/he has sensitivity. In case of sensitivity, the tooth will be deemed to have responded positively to the electrical pulp test and the relevant value will be recorded .If there is no sensitivity, the answer will be accepted as negative.
* Radiographic examination: If swelling, fistula, inflammation or ulceration in the surrounding soft tissue is detected in the visual examination of the relevant tooth, radiological evaluation will be made with periapical radiography. If the patient has a panoramic radiograph obtained in the last 6 months for different treatment needs, it will be used during the clinical examination. Otherwise, a periapical radiograph will be taken from the patient.
* The clinical performance of the restoration will be evaluated with the FDI criteria. Where necessary, digital camera restoration images will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Has to be one of the patients treated with calcium hydroxide as direct pulp capping

Exclusion Criteria:

* Patients (treated with calcium hydroxide as direct pulp capping) who will not be available for the recall appointment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study group consists of a dentist's patients that have been treated with calcium hydroxide as direct pulp capping between 2011-2020.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pulp capping treatment-related adverse events as assessed by vitality tests and intra-oral examination | up to 11 years
  Vitality tests (cold, electrical pulp test) and radiographical examination

SECONDARY OUTCOMES:
Evaluation of the restorations with FDI,World Dental Federation - clinical criteria for the evaluation of direct restorations. | up to 11 years
  The restorations will be evaluated for biological, esthetic and functional parameters as clinically acceptalbe and nonacceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Öztürk Bozkurt, Principal Investigator — fbozkurt@medipol.edu.tr
Locations (1):
- Istanbul Medipol University, Dental School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miles JP, Gluskin AH, Chambers D, Peters OA. Pulp capping with mineral trioxide aggregate (MTA): a retrospective analysis of carious pulp exposures treated by undergraduate dental students. Oper Dent. 2010 Jan-Feb;35(1):20-8. doi: 10.2341/09-038CR1. PMID 20166407
- [Background] Al-Hiyasat AS, Barrieshi-Nusair KM, Al-Omari MA. The radiographic outcomes of direct pulp-capping procedures performed by dental students: a retrospective study. J Am Dent Assoc. 2006 Dec;137(12):1699-705. doi: 10.14219/jada.archive.2006.0116. PMID 17138715